CLINICAL TRIAL: NCT02519530
Title: Multi-site Evaluation of an Evidence-based Positive Youth Development Program: a School-level, Longitudinal, Randomized Controlled Trial
Brief Title: Multi-site Evaluation of an Evidence-based Positive Youth Development Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: Florida Department of Health (Other Government); The Office of Adolescent Health, HHS (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 5 TP1AH000017-04-00
Record Dates: First submitted 2015-07-31; First posted 2015-08-11 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-07

CONDITIONS: Unintended Pregnancy; Adolescent Problem Behavior
Keywords: Positive Youth Development; Teen Outreach; Teen Pregnancy Prevention

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Behavioral: Teen Outreach Program
  Interventions: Behavioral: Teen Outreach Program
- Comparison (No Intervention): This group did not receive TOP, they received business as usual health curriculum offered through the public school system

INTERVENTIONS:
Behavioral: Teen Outreach Program — The Teen Outreach Program (TOP) is a positive youth development program that uses weekly educational peer group sessions, Community Service Learning (CSL), and positive adult guidance to help youth in grades 6-12 build healthy behaviors, life skills, and a sense of purpose. For this study, TOP was implemented in traditional public high schools in Florida and delivered by local health department staff, who were trained and certified as TOP facilitators. Youth enrolled in these classes received the TOP intervention in addition to, not as a replacement for, all business-as-usual curriculum content.
  Arms: Intervention

SUMMARY:
Investigators are carrying out a study to assess the immediate and long-term effects of a positive youth development program (the Teen Outreach Program) on high school youth in Florida. This study will answer the following questions: What is the impact of the Teen Outreach Program on sexual activity and positive youth development at the end of the program and 10 months after the program?

DETAILED DESCRIPTION:
Schools were randomly allocated to either the intervention or the control group. At treatment (intervention) schools, youth participated in TOP in addition to their Health, HOPE, Critical Thinking, Career Research, or Leadership class. At control (non-intervention) schools, youth simply participated in their business-as-usual Health, HOPE, Critical Thinking, Career Research, or Leadership class. Two cohorts of students were recruited for this study, the first cohort joined the study in August 2012 and the second cohort joined the study in August 2013. A survey was given to youth at both treatment and control schools. The paper-and-pencil survey took approximately 30 minutes and asked questions about youth school, grades, peers, health behaviors, and behaviors related to teen pregnancy, including what the participant believes and does in regards to sexual health. The survey was completely confidential and participant names were not linked to survey responses. All survey materials were pre-approved by school administration and the school district office. Participants will be asked to complete the a survey at pre-intervention, post-intervention, and 10-months post-intervention (Cohort 1 only)

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in a class selected for evaluation
* Had parental consent
* Proficient in English
* Capable of independently taking a paper and pencil survey

Exclusion Criteria:

* Not enrolled in a class randomly selected for the evaluation
* They joined a participating class after the completion of the parental consent process
* Not sufficiently proficient in English
* Could not independently take a paper and pencil survey

Ages: 13 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 8161 (Actual)
Dates: Start 2012-08; Primary Completion 2014-10 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Number of participants that report ever having sexual intercourse as measured by the second follow-up youth survey | 10 months post program
  What is the impact of TOP relative to business as usual on ever having sexual intercourse 10 months after the end of the program?
Number of participants that report ever having been pregnant or gotten someone pregnant as measured by the second follow-up youth survey | 10 months post program
  What is the impact of TOP relative to business as usual on ever having been pregnant or gotten someone pregnant 10 months after the end of the program?

SECONDARY OUTCOMES:
Number of participants that report ever having sexual intercourse as measured by the first follow-up youth survey | Immediately post program
  What is the impact of TOP relative to business as usual on ever having sexual intercourse at the end of the program?
Number of participants that report ever having been pregnant or gotten someone pregnant as measured by the first follow-up youth survey | Immediately post program
  What is the impact of TOP relative to business as usual on ever having been pregnant or gotten someone pregnant at the end of the program?

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Daley, Ph.D, Principal Investigator — University of South Florida; Eric Buhi, Ph.D, Principal Investigator — San Diego State University

REFERENCES:
- [Derived] Marhefka SL, Noble CA, Walsh-Buhi ER, Turner D, Mahony H, Singleton A, DeBate R, Daley EM. Key Considerations and Recommended Strategies for Conducting a School-Based Longitudinal RE-AIM Evaluation: Insights From a 28-School Cluster Randomized Trial. Health Promot Pract. 2023 Jan;24(1):160-171. doi: 10.1177/15248399211042339. Epub 2021 Oct 4. PMID 34605711
- [Derived] Walsh-Buhi ER, Marhefka SL, Wang W, Debate R, Perrin K, Singleton A, Noble CA, Rahman S, Maness SB, Mahony H, Ziemba R, Malmi M, Marwah E, Hall K, Turner D, Blunt-Vinti H, Noble SM, Daley EM. The Impact of the Teen Outreach Program on Sexual Intentions and Behaviors. J Adolesc Health. 2016 Sep;59(3):283-290. doi: 10.1016/j.jadohealth.2016.05.007. Epub 2016 Jun 16. PMID 27318427